CLINICAL TRIAL: NCT03671460
Title: Phase I Study of the Safety and Efficacy of CD19 CAR-T Cells in Patients With Relapsed or Refractory Acute B-cell Lymphoblastic Leukemia (R/R B-ALL)
Brief Title: CD19 CAR-T Cells for Patients With Relapse and Refractory CD19+ B-ALL.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Mycure Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TianjinMycure-LDP-CD19 CAR-T
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: B-cell acute lymphoblastic leukemia; CD19 CAR-T
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Intervention Model Description: single-center, open-label, nonrandomized, no control, prospective clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-CAR-T Cells (Experimental): Subjects will receive CD19-CAR-T Cells on Day 0 : 100% of total dose.
  Interventions: Biological: CD19 CAR-T cells

INTERVENTIONS:
Biological: CD19 CAR-T cells — T cells purified from the PBMC of subjects, transduced with 4-1BB/CD3-ζ lentiviral vector, expanded in vitro for future administration.

SUMMARY:
This is a single center, single arm, open-lable phase 1 study to determine the safety and efficacy of CD19-CAR-T cells in patients with relapsed or refractory acute B-cell lymphoblastic leukemia (R/R B-ALL).

DETAILED DESCRIPTION:
In this single-center, open-label, nonrandomized, no control, prospective clinical trial, no less than 18 CD19+ B-cell relapsed or refractory acute B-cell lymphoblastic leukemia (R/R B-ALL) patients will be enrolled. Side effects of CD19 CAR T cells therapy will be monitored. The purpose of current study is to determine the clinical efficacy and safety of CD19 CAR T cells therapy in patients with R/R B-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. More than 1 year;
2. CD19 positive B-cell acute lymphoblastic leukemia;
3. Important organ function is satisfied: cardiac ultrasound indicates cardiac ejection fraction ≥50%, no obvious abnormality in ECG; blood oxygen saturation ≥90%; creatinine clearance calculated by Cockcroft-Gault formula ≥40ml/min; ALT and AST≤ 5 times normal range, total bilirubin ≤ 34.2 μmol / L.
4. Expected to survive for more than 3 months;
5. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. Recent or current use of glucocorticoid or other immunosuppressor;
2. Uncontrolled active infection, HIV infection, syphilis serology reaction positive;
3. Has a graft-versus-host response and requires the use of immunosuppressants；
4. Drug uncontrollable central nervous system leukemia；
5. Pregnant or lactating female；
6. The patient did not agree to use effective contraception during the treatment period and for the following 1 year；
7. A history of other malignant tumors;
8. The investigator believes that there are other factors that are not suitable for inclusion or influence the subject's participation or completion of the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-09-07 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events | 6 months
  Percentage of participants with adverse events

SECONDARY OUTCOMES:
complete remission rate | 6 months
  The percentage of participants who achieved complete remission (CR) over all participants (CRR).
objective remission rate | 6 months
  The percentage of participants who achieved complete remission (CR) and partial remission over all participants (ORR).

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD,MD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided
We don't decide when to share IPD and what will be shared.